CLINICAL TRIAL: NCT01761136
Title: Phase 4 Study of Haemophilus Influenzae Type b Vaccine in Different Injection Site
Brief Title: The Safety and Immunogenicity of Haemophilus Influenzae Type b Vaccine in Different Injection Site
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BJCDPC-4
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
MeSH Terms: interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inoculation in upper arm deltoid (Active Comparator): Inoculation of Hib vaccine of two brands in upper arm deltoid
  Interventions: Biological: Inoculation in upper arm deltoid; Biological: Inoculation in vastus lateralis muscle
- Inoculation in vastus lateralis muscle (Experimental): Inoculation of Hib vaccine of two brands in vastus lateralis muscle
  Interventions: Biological: Inoculation in upper arm deltoid; Biological: Inoculation in vastus lateralis muscle

INTERVENTIONS:
Biological: Inoculation in upper arm deltoid — Inoculation of Hib vaccine of two brands in upper arm deltoid
Biological: Inoculation in vastus lateralis muscle — Inoculation of Hib vaccine of two brands in vastus lateralis muscle

SUMMARY:
The objective of this study was to evaluate the safety and immunogenicity of Haemophilus influenzae type b vaccine in different injection site.

DETAILED DESCRIPTION:
A randomized trial was conducted in 680 healthy infants with Hib vaccine of two brands. The different sub-groups were selected randomly based on the plan to inoculate vaccines in the upper arm deltoid or vastus lateralis muscle. The safety and immunogenicity were assessed after three or two doses.

ELIGIBILITY:
Inclusion Criteria:

* participants were under 1 years old, and were in good healthy
* participants were full-time pregnancy and birth weight were more than 2.5 kg

Exclusion Criteria:

* current infectious fever or acute disease
* a history of hypersensitivity to study vaccine components especially tetanus toxoid
* a history of allergy, autoimmune, convulsions, seizures heredity disease
* a history of Hib vaccination or Hib disease
* a history of congenital deformity, developmental disorders or serious chronic diseases, muscle injection contradiction, and immunosuppressive agents, hormone or immunoglobulin received.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 680 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse events of Haemophilus influenzae type b vaccine in different injection site | one year

SECONDARY OUTCOMES:
Antibody titre of Haemophilus influenzae type b vaccine in different injection site | one year

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Principal Investigator — Beijing Chaoyang District Center for Disease Control and Prevention
Locations (5):
- China (5):
  - Beijing Huaxin Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Women's and Children's Hospital, Beijing
  - Beijing Dongba Hospital, Beijing
  - Cuigezhuang community health service centers, Beijing
  - Xiaohongmen community health service centers, Beijing